CLINICAL TRIAL: NCT03443934
Title: Hemodynamic Alterations in Liver Cirrhosis Compared to Healthy Subjects: Assessment of Non-invasive MRI and Echocardiography Compared to Liver Vein Catheterization
Brief Title: Hemodynamic Alterations in Liver Cirrhosis Validated by Non-invasive MR Compared to Invasive Assessment
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Flemming Bendtsen, Professor, MD, Hvidovre University Hospital
Other Study IDs: 16048555
Record Dates: First submitted 2018-02-10; First posted 2018-02-23 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Portal Hypertension; Liver Diseases; Liver Cirrhoses; Cirrhosis
Keywords: Hemodynamic assessments; Echocardiography; MR-Elastography; Liver vein catheterization; Liver Cirrhosis; Cirrhotic cardiomyopathy; Cirrhotic complications; Magnetic Resonance Imaging
MeSH Terms: conditions — Hypertension, Portal; Liver Diseases; Fibrosis; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Standard clinical blood tests and pertinent bioactive substances is measured in blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver cirrhosis is a chronic disease characterized by a progressive accumulation of fibrosis, loss of liver function and portal hypertension leading to several hemodynamic changes.The exact pathophysiological mechanisms causing the hyperdynamic alterations in cirrhosis are not fully elucidated.

Aim:

The aim of the study is to assess hemodynamic alterations in liver cirrhosis by non-invasive MRI and echocardiography compared to portal hypertension measured with liver vein catheterization (HVPG, hepatic vein pressure gradient). Furthermore, the aim is to explore hemodynamic differences between cirrhotic patients and healthy subjects.

Study design and cohort:

The study has a cross-sectional design and a cohort with 99 patients with liver cirrhosis - with and without complications and 27 healthy volunteers. The patients are recruited at the Gastrounit Hvidovre University Hospital.

The day before the first visit patients are hospitalized and fasting overnight. At first visit liver vein catheterization (LVC) and echocardiography are performed. Second visit must be performed within 4 weeks after first visit. At the second visit patients are fasting minimum 6 hours before having MR-flow scanning, cardiac-MR and MR-Elastography (MR-E).

The healthy volunteers are only offered MR-flow scanning, cardiac MR and MR-E as well as urine- and blood tests

Follow-up for liver-related clinical outcome and mortality in medical records

DETAILED DESCRIPTION:
MR elastography, cardiac scan, phase contrast MRI of blood flow compared to LVC

ELIGIBILITY:
Inclusion Criteria:

Patients with liver cirrhosis or portal hypertension Patient of more than 18 and less than 82 years of age

Exclusion Criteria:

Patients who are unable to give informed consent Patients with absolute contraindication for MRI Pregnant women Patient with severe hemodynamic comorbidity

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort with 99 cirrhotic patients with and without complications and 27 healthy volunteers. The patients are recruited at the Gastrounit Hvidovre University Hospital
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
MRI-flow (mL/min) in splanchnic arterial compared to clinical severity of cirrhosis and to portal hypertension measured as HVPG (mmHg) during liver vein catheterization | During MRI-scan
  To compare the flow and cardiac parameters measured by MRI with disease progression and with HVPG (mmHg) measured during liver vein catheterization (LVC)

SECONDARY OUTCOMES:
Hemodynamic alterations in patients with liver cirrhosis measured as flow (mL/min) in relevant vessels compared to flow in healthy subjects | During MRI-scan
  To characterize flow in cirrhotic patients compared to healthy subjects
Measurements of hemodynamic alterations compared with different severity of liver cirrhosis defined by Child Pugh and MELD score | During MRI-scan
  To assess the relation between severity of cirrhosis with changes in flow and cardiac-MRI
MR-elastography measurements (kPa) to characterize severity of cirrhosis categorized with Child Pugh, MELD and HVPG | During MRI-scan
  To assess the relation between severity of cirrhosis and changes in liver and spleen stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Bendtsen, Professor, Principal Investigator — Professor
Locations (1):
- Centre of Gastroenterology, Dept. of medicine. Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mynster Kronborg T, Webel H, O'Connell MB, Danielsen KV, Hobolth L, Moller S, Jensen RT, Bendtsen F, Hansen T, Rasmussen S, Juel HB, Kimer N. Markers of inflammation predict survival in newly diagnosed cirrhosis: a prospective registry study. Sci Rep. 2023 Nov 16;13(1):20039. doi: 10.1038/s41598-023-47384-2. PMID 37973887
- [Derived] Danielsen KV, Wiese S, Busk T, Nabilou P, Kronborg TM, Petersen CL, Hove JD, Moller S, Bendtsen F. Cardiovascular Mapping in Cirrhosis From the Compensated Stage to Hepatorenal Syndrome: A Magnetic Resonance Study. Am J Gastroenterol. 2022 Aug 1;117(8):1269-1278. doi: 10.14309/ajg.0000000000001847. Epub 2022 Jun 3. PMID 35916685